CLINICAL TRIAL: NCT04214769
Title: Evaluation of the Effect of Radiation Therapy Among Head and Neck Cancer Patients on the Inner Ear Function Using Novel Techniques
Brief Title: Effect of Radiation Therapy Among Head and Neck Cancer Patients on the Inner Ear Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 403-19
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Cancer Patients Treated With Radiotherapy
MeSH Terms: interventions — Audiometry; Acoustic Impedance Tests; Electronystagmography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancer patients
  Interventions: Diagnostic Test: Audiometry and tympanometry, vHIT, VEMP, ENG

INTERVENTIONS:
Diagnostic Test: Audiometry and tympanometry, vHIT, VEMP, ENG — Diagnostic tests

SUMMARY:
Aims: 1. To evaluate the effects of radiation therapy on the inner ear, among patients treated with radiation therapy for head and neck cancers using a wide battery of tests (Audiometry and tympanometry, vHIT, VEMP, ENG) ; 2. To correlate the mean total radiation dose to the cochlea with the effects on audiological and vestibular function

ELIGIBILITY:
Inclusion Criteria:

* Females and males, Age: ≥ 18 years old
* Patients diagnosed Head and Neck cancers, not treated previously
* Planned for radiation therapy in which the inner ear will be radiated

Exclusion Criteria:

* Patients who were previously diagnosed with a vestibular disorder
* Previous middle or inner ear anomaly
* Failure to complete the whole course of radiation therapy
* More than one course of radiation therapy
* Patients treated with concurrent ototoxic chemotherapy
* Pregnant women
* Patients who will not sign an informed consent form
* Helpless or incompetent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed Head and Neck cancers, not treated previously, and planned for radiation therapy in which the inner ear will be radiated
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Audiometry | 1.5 Year
  The change in hearing threshold and in the speech-audiometry
ENG test | 1.5 Year
  Abnormal function of the central vestibular pathways, unilateral weakness of the vestibular apparatus or direction preponderance
VEMP test | 1.5 Year
  Abnormal latencies, amplitudes, thresholds
vHIT test | 1.5 Year
  abnormal gain, the appearance of overt and covert saccades

IPD SHARING:
Plan to Share IPD: No